CLINICAL TRIAL: NCT04530825
Title: Addressing Social Determinants of Health During Clinical Care Visits to Promote Equitable Behavior Change and PREVENT Cardiovascular Disease
Brief Title: PREVENT Tool Study: Late Effects Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202007026; K12HL137942 (NIH)
Record Dates: First submitted 2020-08-11; First posted 2020-08-28 (Actual); Results first posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Cardiovascular Disease; Childhood Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Providers (No Intervention): * All eligible providers will be sent questionnaires electronically to their email at baseline and follow-up. Providers will be invited to attend a training session to educate them on the PREVENT tool at baseline
  * A subset of 5-10 providers will be recruited via email, at the baseline training,or by using snowball-sampling approach within the clinic to participate in qualitative in-depth interviews
- Parents (No Intervention): -Semi-structured interviews
- Patients - Wait-List Control (Active Comparator): * Complete questionnaires at baseline (administered electronically or by mail; accelerometers administered by mail). Following baseline measurement, patients will be randomized and attend their clinic visit. Follow-up measures will be administered immediately following the clinic visit (within 48 hours) and 3-months after the clinic visit electronically and by mail
  * Up to 10 patients will also take part in semi-structured interviews
  * A PREVENT action plan (behavior change prescription, community resources, and education) will be provided to the patient via email after the completion of the follow-up measurement.
  Interventions: Other: Wait-List Control
- Patients - PREVENT tool (Experimental): * Complete questionnaires at baseline (administered electronically or by mail; accelerometers administered by mail). Following baseline measurement, patients will be randomized and attend their clinic visit. Follow-up measures will be administered immediately following the clinic visit (within 48 hours) and 3-months after the clinic visit electronically and by mail
  * Up to 10 patients will also take part in semi-structured interviews
  * At the clinic visit, the provider will use PREVENT tool to discuss risk and deliver a tailored behavioral change plan inclusive of patient-centered community resources. PREVENT will calculate patient's overall risk for developing cardiovascular disease. Physical activity and food intake recommendations are tailored to current weight status and health behaviors using evidence-based recommendations.
  Interventions: Other: PREVENT Tool

INTERVENTIONS:
Other: Wait-List Control — -Will receive routine clinical care. After completion of follow-up measures, control participants will receive a behavior change prescription via the PREVENT tool
  Arms: Patients - Wait-List Control
Other: PREVENT Tool — -PREVENT is a novel Health Information Technology tool designed to promote physical activity and healthy food intake among overweight/obese adolescent patients at the point of care. PREVENT automates the delivery of personalized, evidence-based behavior change recommendations and provides an interactive map of community resources to help providers link patients to resources in their community.
  Arms: Patients - PREVENT tool

SUMMARY:
The purpose of this study is to test the feasibility of a novel, Health Information Technology behavior change tool in a single clinic setting. The PREVENT tool is the first electronic health record (EHR)-compatible tool that both tailors evidence-based behavior change strategies and incorporates community-level data specific to each patient into routine care. The central hypothesis is that PREVENT will improve patient's attitudes towards behavior change recommendations, increase adherence to recommended behavior change and improve cardiovascular health. Fifty adolescents will be randomized to intervention or wait-list, routine care control to assess the preliminary effectiveness of PREVENT. Qualitative and quantitative methods will be used among patients, parents and providers to examine barriers to current and future implementation of the PREVENT tool to inform adoption and maintenance.

ELIGIBILITY:
Inclusion Criteria:

Patient Eligibility Criteria:

* Adolescents 12 to 19 years
* Prior diagnosis of pediatric cancer (diagnosed <21 years of age)
* Not receiving active therapy for their cancer
* Receiving care from the Pediatric Hematology/Oncology staff and physicians at St. Louis Children's Hospital or the St. Louis Children's Specialty Care Center (CSCC)
* At risk for poor cardiovascular health (CVH) (BMI greater than or equal to 85th percentile)

Provider Eligibility Criteria -All providers and staff (physicians, nurses, clinic staff, clinical research associates) in the Pediatric Hematology/Oncology program at St. Louis Children's Hospital and the CSCC

Parent Eligibility Criteria

-A parent or legal guardian of a study participant. The parent or legal guardian must have been present at the clinic visit in which the PREVENT tool was administered to the study participant.

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maura Kepper, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Providers: * All eligible providers were sent questionnaires electronically to their email at baseline and follow-up. Providers were invited to attend a training session to educate them on the PREVENT tool at baseline
  * A subset of 5-10 providers were recruited via email, at the baseline training, or by using snowball-sampling approach within the clinic to participate in qualitative in-depth interviews
- Patients - Wait-List Control: * Completed questionnaires at baseline (administered electronically or by mail; accelerometers administered by mail). Following baseline measurement, patients were randomized and attended their clinic visit. Follow-up measures were administered immediately following the clinic visit (within 48 hours) and 3-months after the clinic visit electronically and by mail
  * Up to 10 patients took part in semi-structured interviews
  * A PREVENT action plan (behavior change prescription, community resources, and education) was provided to the patient via email after the completion of the follow-up measurement.
- Patients - PREVENT Tool: * Completed questionnaires at baseline (administered electronically or by mail; accelerometers administered by mail). Following baseline measurement, patients were randomized and attended their clinic visit. Follow-up measures were administered immediately following the clinic visit (within 48 hours) and 3-months after the clinic visit electronically and by mail
  * Up to 10 patients took part in semi-structured interviews
  * At the clinic visit, the provider used the PREVENT tool to discuss risk and deliver a tailored behavioral change plan inclusive of patient-centered community resources. PREVENT calculates patient's overall risk for developing cardiovascular disease. Physical activity and food intake recommendations are tailored to current weight status and health behaviors using evidence-based recommendations.
Period: Overall Study
Arm/Group | Providers | Parents | Patients - Wait-List Control | Patients - PREVENT Tool
Started | 7 | 29 | 16 | 13
Completed | 4 | 28 | 16 | 12
Not Completed | 3 | 1 | 0 | 1
Not completed — No longer eligible on the day of baseline visit | 0 | 1 | 0 | 1
Not completed — Did not complete follow-up | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Providers | Parents | Patients - Wait-List Control | Patients - PREVENT Tool | Total
Number analyzed (Participants) | 4 | 28 | 16 | 12 | 60
Age, Continuous [Median (Full Range); unit: years] — Population: Age was not collected on Parents.
  years
    number analyzed (Participants) | 4 | 0 | 16 | 12 | 32
    (all) | 40.5 [36 to 62] |  | 16.0 [13 to 19] | 17.0 [12 to 19] | 19.4 [12 to 62]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex was not collected on Parents.
  Participants
    number analyzed (Participants) | 4 | 0 | 16 | 12 | 32
    Female | 3 |  | 6 | 6 | 15
    Male | 1 |  | 10 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity was not collected on Parents.
  Participants
    number analyzed (Participants) | 4 | 0 | 16 | 12 | 32
    Hispanic or Latino | 0 |  | 0 | 0 | 0
    Not Hispanic or Latino | 4 |  | 16 | 12 | 32
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race was not collected on Parents.
  Participants
    number analyzed (Participants) | 4 | 0 | 16 | 12 | 32
    American Indian or Alaska Native | 0 |  | 0 | 0 | 0
    Asian | 1 |  | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0 | 0
    Black or African American | 0 |  | 0 | 1 | 1
    White | 3 |  | 15 | 9 | 27
    More than one race | 0 |  | 1 | 2 | 3
    Unknown or Not Reported | 0 |  | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 28 | 16 | 12 | 60

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Minutes of Moderate Physical Activity Per Week (From Self Report) Survey
Description: * Physical activity will be measured using a triaxial accelerometer (Actigraph GT3X+, Actigraph of Ft. Walton Beach, FL). The participant will be instructed to wear the accelerometer on an elasticized belt, on the left mid-axillary line. The Actigraph is one of the most common accelerometers used for scientific purposes. Participants will be encouraged to wear the accelerometer 24-hours per day for at least 7-days, including 2 weekend days. Participants completed a brief Health Behavior & Attitudes Survey using questions from the International Physical Activity Questionnaire Mean changes from baseline and 3-month follow-up were calculated as the follow-up measure minus the baseline measure, averaged across the intervention groups.
  * Note: Actigraph measure was dropped due to university mail distribution delays during the remote work period of the COVID-19 pandemic. Self-reported change in minutes of physical activity became the primary outcome.
Time Frame: At baseline and 3-months
Population: Providers and parents were not evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | Providers | Parents | Patients - Wait-List Control | Patients - PREVENT Tool
Number analyzed (Participants) | 0 | 0 | 16 | 12
minutes/week |  |  | 43.3 (341.6) | 16.8 (357.7)

2. Primary Outcome: Mean Change in Minutes of Vigorous Physical Activity Per Week (From Self Report) Survey
Description: as for outcome 1
Time Frame: At baseline and 3-months
Population: Providers and parents were not evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | Providers | Parents | Patients - Wait-List Control | Patients - PREVENT Tool
Number analyzed (Participants) | 0 | 0 | 16 | 12
minutes/week |  |  | -211.4 (241.6) | -1.4 (109.0)

3. Primary Outcome: Mean Change in Number of Food Intake Behaviors Met
Description: Patient-reported food intake behaviors (fruit and vegetable intake, whole grains, sugar-sweetened beverages and snacking behaviors) are collected using a brief Health Behavior & Attitudes Survey. Responses are dichotomized into a binary yes (1)/no (0) score indicating whether or not the patient is meeting the food intake recommendation for each food group. The total number of food intake behaviors are scored on a 5 item scale (range 0-5), maximum improvement in number of behaviors=5. Mean changes from baseline and 3-month follow-up were calculated as the follow-up measure minus the baseline measure, averaged across the intervention groups.
Time Frame: At baseline and 3-months
Population: Providers and parents were not evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a 0-5 scale
Arm/Group | Providers | Parents | Patients - Wait-List Control | Patients - PREVENT Tool
Number analyzed (Participants) | 0 | 0 | 16 | 12
score on a 0-5 scale |  |  | 0.15 (1.1) | 0.78 (1.9)

4. Primary Outcome: Provider's Satisfaction of PREVENT Tool: Survey
Description: A survey (24-questions) containing validated subscales assessed provider's satisfaction with the PREVENT tool on subscales assessing acceptability, feasibility, and appropriateness of the tool, and satisfaction with specific components of the tool. Items were scored on a 5-point Likert scale with a higher score indicating greater satisfaction. Subscales were summed to generate the average across all questions (range 1-5) and was reported as overall satisfaction.
Time Frame: 3-months
Population: Parents and patients were not evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Providers | Parents | Patients - Wait-List Control | Patients - PREVENT Tool
Number analyzed (Participants) | 4 | 0 | 0 | 0
score on a scale | 3.61 (1.1) |  |  |

5. Primary Outcome: Fidelity of PREVENT Tool Implementation
Description: Fidelity will be measured using direct observation of patient-provider interactions while using the PREVENT tool. A direct observation checklist will be used by the observer to determine the number of interactions with the PREVENT tool that were implemented as intended.
Time Frame: 0-3 months
Population: Data was not collected on this outcome measure as the study team was unable to consistently observe study visits due to COVID-19 restrictions.
Arm/Group | Providers | Parents | Patients - Wait-List Control | Patients - PREVENT Tool
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Provider's Motivation for Sustained Use of PREVENT Tool
Description: A survey (8 questions) assessed provider's intent to change their behavior and continue using PREVENT. Questions were adapted from Legare's CPD Reaction Questionnaire and asked using a 5-point Likert scale (range 1-5). An average of all responses was calculated with a higher score indicating greater motivation for sustained use.
Time Frame: 3-months
Population: Parents and patients were not evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Providers | Parents | Patients - Wait-List Control | Patients - PREVENT Tool
Number analyzed (Participants) | 4 | 0 | 0 | 0
score on a scale | 2.79 (1.2) |  |  |

7. Secondary Outcome: Maintenance of PREVENT Tool as Measured by Provider Perceptions of Feasibility of the Tool
Description: Qualitative in-depth interview with providers who used the PREVENT tool. Qualitative content analysis methods were used to summarize key themes related to provider perceptions of the tool and ability to use the tool in routine clinical practice.
Time Frame: 3-months
Population: Parents and patients were not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Providers | Parents | Patients - Wait-List Control | Patients - PREVENT Tool
Number analyzed (Participants) | 4 | 0 | 0 | 0
Participants
  More feasible to deliver PREVENT during longer appointments; time could be a barrier | 4 |  |  |
  More feasible to have clinic staff that could prepare the tool and review recommendations | 4 |  |  |
  Lack of electronic health record integration was a key barrier to using PREVENT in routine practice. | 4 |  |  |

8. Secondary Outcome: Maintenance of PREVENT Tool as Measured by Provider Perceptions of Ease of Use of the Tool
Description: as for outcome 7
Time Frame: 3-months
Population: Parents and patients were not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Providers | Parents | Patients - Wait-List Control | Patients - PREVENT Tool
Number analyzed (Participants) | 4 | 0 | 0 | 0
Participants
  User friendly, easily navigable platform; color coding and visualizations were easy to understand | 4 |  |  |
  Providers liked having clear, concrete recommendations to give patients | 4 |  |  |

9. Secondary Outcome: Patient's Perceptions of Usability/Acceptability of PREVENT Tool
Description: Semi-structured interviews with adolescent study participants (n=10).
Time Frame: 3-months
Population: Data was not collected on this outcome measure as the investigators were unable to successfully recruit patients for follow-up interviews over the phone.
Arm/Group | Providers | Parents | Patients - Wait-List Control | Patients - PREVENT Tool
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Parent's Perceptions of Usability/Acceptability of PREVENT Tool
Description: Semi-structured interviews with parents/guardians (n=10) of study participants.
Time Frame: 3-months
Population: Data was not collected for this outcome measure as the investigators were unable to successfully recruit parents for follow-up interviews over the phone.
Arm/Group | Providers | Parents | Patients - Wait-List Control | Patients - PREVENT Tool
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Impact of PREVENT Tool on Mean Change in Patient's Body Mass Index (BMI)
Description: Collected from patient's medical record. BMI z-score is a standardized calculation accounting age and sex using the Centers for Disease Control and Prevention Growth Charts. A z-score represents the standard deviation from the population mean. A z-score of zero represents the population mean. Mean change in BMI z-score was calculated by subtracting the baseline mean from the follow-up mean for each intervention group. A decrease in z-score is a favorable outcome.
Time Frame: At baseline and 3-months
Population: Parents and providers were not evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Providers | Parents | Patients - Wait-List Control | Patients - PREVENT Tool
Number analyzed (Participants) | 0 | 0 | 16 | 12
z-score |  |  | 0.09 (0.22) | -.03 (0.16)

12. Secondary Outcome: Impact of PREVENT Tool on Patient's Systolic and Diastolic Blood Pressure
Description: Collected from patient's medical record. Blood pressure is measured in mmHg. The mean change was calculated by subtracting the baseline mean from the follow-up mean for each intervention group.
Time Frame: At baseline and 3-months
Population: Parents and providers were not evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Providers | Parents | Patients - Wait-List Control | Patients - PREVENT Tool
Number analyzed (Participants) | 0 | 0 | 16 | 12
mmHg
  Systolic blood pressure |  |  | -1.38 (10.0) | 0.65 (11.1)
  Diastolic blood pressure |  |  | -0.49 (6.7) | -1.83 (10.5)

13. Secondary Outcome: Impact of PREVENT Tool on Patient's Cholesterol
Description: Collected from patient's medical record
Time Frame: At baseline and 3-months
Population: Data was not collected and outcome measure was dropped.
Arm/Group | Providers | Parents | Patients - Wait-List Control | Patients - PREVENT Tool
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Impact of PREVENT Tool on Patient's Fasting Blood Glucose
Description: Collected from patient's medical record
Time Frame: At baseline and 3-months
Population: Data was not collected and outcome measure was dropped.
Arm/Group | Providers | Parents | Patients - Wait-List Control | Patients - PREVENT Tool
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Impact of PREVENT Tool on Patient's Attitudes Toward Behavior Change
Description: A survey (6-question) administered to patients will assess attitudes toward and readiness for behavior change. Questions are asked using a 5-point Likert scale (range: 0-5) with a higher score indicating more positive attitudes.
Time Frame: At baseline and 3-months
Population: Parents and providers were not evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Providers | Parents | Patients - Wait-List Control | Patients - PREVENT Tool
Number analyzed (Participants) | 0 | 0 | 16 | 12
score on a scale |  |  | 0.16 (0.76) | 0.23 (1.08)

16. Secondary Outcome: Clinic-level Capacity for Sustainability as Measured by Provider Survey
Description: The Clinical Sustainability Assessment Tool (CSAT) will assess clinic-level readiness and capacity for sustainability of the PREVENT tool. The CSAT tool will examine organization, financial, regulatory and political factors that may influence sustainability. 10 items scored on a 7-point scale, with higher scores indicating greater capacity for sustainment. The average of the 10 items is reported (range 1-7).
Time Frame: 3-months
Population: Parents and patients were not evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Providers | Parents | Patients - Wait-List Control | Patients - PREVENT Tool
Number analyzed (Participants) | 4 | 0 | 0 | 0
score on a scale | 3.63 (2.03) |  |  |

ADVERSE EVENTS:
Time Frame: From baseline through 6 months post-baseline.
Description: Adverse events and all-cause mortality were not collected for providers or parents.
Arm/Group | Providers | Parents | Patients - Wait-List Control | Patients - PREVENT Tool
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/16 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/16 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT04530825/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/25/NCT04530825/ICF_001.pdf